CLINICAL TRIAL: NCT03420820
Title: Concentrating on Antisepsis: 5% vs. 10% Povidone-Iodine Prior to Intravitreal Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Matthew Bolton (Other)
Responsible Party: Sponsor-Investigator, Matthew Bolton, Ophthalmology Resident, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1162018
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Endophthalmitis; Eye Infections
Keywords: intravitreal injection; povidone-iodine; ocular surface flora; endophthalmitis; betadine
MeSH Terms: conditions — Endophthalmitis; Eye Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5% Betadine, Ocular Surface only (Experimental): Use of 5% P-I from bottle dropper to sterilize the ocular surface only, prior to injection. Intervention: bacterial culture swab.
  Interventions: Biological: Bacterial Culture Swab
- 10% Betadine, Ocular Surface only (Experimental): Use of 10% P-I swabstick to sterilize the ocular surface only, prior to injection. Intervention: bacterial culture swab.
  Interventions: Biological: Bacterial Culture Swab
- 10% Betadine, Ocular Surface and Adnexa (Experimental): Use of 10% P-I swabstick to sterilize the ocular surface and surrounding lids and eyelashes only, prior to injection. Intervention: bacterial culture swab.
  Interventions: Biological: Bacterial Culture Swab

INTERVENTIONS:
Biological: Bacterial Culture Swab — Culture swabs will be obtained before application of PI and after injection.

SUMMARY:
This is a randomized controlled single blind prospective study evaluating the efficacy of ocular surface sterilization between three different povidone-iodine preparation techniques prior to intravitreal injection. The primary end point is significant different between median colony-forming units pre- and post-sterilization and injection.

DETAILED DESCRIPTION:
Introduction: An estimated 5.9 - 7.9 million intravitreal injections (IVI) were given in 2016. While the incidence of post-injection endophthalmitis is exceedingly low, it is a feared complication of the procedure. 96% of culture-positive post-injection endophthalmitis cases are caused by conjunctival commensals, emphasizing the importance of ocular surface sterilization prior to IVI. The most recently published guidelines for IVI state that "Povidone-Iodine (5-10%) should be the last agent applied to the intended injection site before the injection," a recommendation that is universally followed. However, there is no standard of care regarding the concentration of PI nor the field of sterilization (e.g, cleaning the eyelids and lashes), and technique varies widely in clinical practice. The literature reveals no direct comparison of 5% vs 10% PI in the context of intravitreal injection.

Methods: Single-center randomized prospective trial enrolling patients into three protocols: 5% P-I applied to ocular surface from bottle, 10% P-I swabstick applied to ocular surface, and 10% P-I swabstick applied to lids, lashes, and ocular surface. Pre-procedure cultures will be obtained from the ocular surface, and a second culture will be taken following antisepsis, injection, and irrigation. Standard microbiologic techniques will be used to collect, culture, identify, and quantify ocular surface bacteria counts. Kruskal Wallis test will be used to assess significant difference between median bacterial loads at baseline and post-cleaning, as well as median reduction from baseline. Chi-squared test will be used to assess significant difference between reduction in number of patients with specific bacteria. Following injection, a patient survey will be administered to compare patients' subjective symptoms of ocular surface irritation during the PI preparation phase of the procedure.

Conclusions: The investigators anticipate that no significant difference exists in decrease of median CFUs between the three protocols, and that lower concentration of P-I provides a more comfortable patient experience.

ELIGIBILITY:
Inclusion Criteria:

* enrollment will be open to men and women of all ethnic backgrounds between the ages of 18-100 who are offered intravitreal injections by Dr. Anthony Mazzulla at his Retina clinic at the Ochsner Clinic Foundation as a treatment for diabetic macular edema, proliferative diabetic retinopathy, age related exudative macular degeneration, or any other cause of choroidal neovascularization or cystoid macular edema.

Exclusion Criteria:

* Current eye infection, actively treated blepharitis, current use of topical or systemic antimicrobial agents, current use of topical or systemic corticosteroids, allergy to iodine, pregnancy, children.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Median Colony-Forming Units | 3 months
  Median CFUs compared pre- and post-injection

SECONDARY OUTCOMES:
Patient's ocular surface symptoms during sterilization with povidone-iodine | 3 months
  Survey-based

CONTACTS AND LOCATIONS:
Overall Officials: Donald Mazzulla, MD, Principal Investigator — Ochsner Health System

IPD SHARING:
Plan to Share IPD: No